CLINICAL TRIAL: NCT00536796
Title: Non-interventional Study Investigating How Effective Secondary Prevention Patients Are Treated to Their LDL-C Targets
Brief Title: Percentage of Secondary Prevention Patients Treated to Their LDL-C Targets
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CAT-CRE-2007/2
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Hyperlipidemias; Atherosclerosis; Coronary Heart Disease; Carotid Stenosis; Peripheral Vascular Diseases; Diabetes Mellitus
Keywords: Hyperlipidemia; Need-to-treat; NIS; Secondary prevention patients with hyperlipidemia and atherosclerosis (coronary heart disease, carotid stenosis, PVD, etc.) and/or diabetes
MeSH Terms: conditions — Hyperlipidemias; Atherosclerosis; Coronary Disease; Carotid Stenosis; Peripheral Vascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Patients at very high risk
- Patients at high risk
- Patients at medium risk
- Patients at low risk

SUMMARY:
A cholesterol/lipid profile screening project of high risk patients with hyperlipidaemia (secondary prevention) who already receive cholesterol-lowering therapy. Lipid profile and rate of patients who are treated to target (which is <100mg/dl for patients with high risk and <70mg/dl for patients at very high risk) are screened (hospital-based specialists). The doctors therapy decisions after the screening and possible reasons for these decisions will be documented. Our aim is to evaluate dosing habits, to evaluate how many patients are treated to their LDL-C target and to underline the importance of treating patients to their cholesterol targets.

ELIGIBILITY:
Inclusion Criteria:

* Secondary prevention patients with hyperlipidemia and atherosclerosis (coronary heart disease, carotid stenosis, PVD, etc.) and/or diabetes who already receive cholesterol-lowering therapy

Exclusion Criteria:

* Patients who do not receive cholesterol-lowering therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female secondary prevention patients with: coronary disease with event: acute coronary syndrome, status post MI, PTCA, CABG, angiographically verified), PAVK (min. IIb or S.p. revascularization), stroke/TIA, carotis-plaque (asymptomatic min. 70% or S.p. revascularization), Diabetes Mellitus (type I, II)
Sampling Method: Non-Probability Sample
Enrollment: 1096 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cholesterol levels | After 4 weeks
  Cholesterol levels from high risk patients after 4 weeks of cholesterol-lowering drug therapy under target values

CONTACTS AND LOCATIONS:
Overall Officials: Josef Patsch, MD, Study Chair — Chair of the Austrian Atheroslerosis Society; Bernhard Foger, MD, Study Chair — Co-Chair of the Austrian Atheroslerosis Society
Locations (1):
- Research Site, Rohrbach, Upper Austria, Austria